CLINICAL TRIAL: NCT05368948
Title: The Assessment of Antimicrobial Peptides Against Fungal Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara salah abd El mawgoud, Assistant lecturer in clinical pathology department, Assiut University
Other Study IDs: antimicrobial peptides
Record Dates: First submitted 2022-04-14; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Fungal Infection
Keywords: antimicrobial peptides
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Identification of different types of fungi.
* Determine sensitivity the profile and the resistance pattern of the clinical isolates against antifungal.
* Determine the antifungal effects of defensin, cathelicidin and histatins and their effects on biofilm formation and resistant isolates.

DETAILED DESCRIPTION:
Fungal infections are recurrent in the clinical environment and, annually, affect 25% of the general population worldwide, causing high morbidity and mortality rates. The indiscriminate use of broad-spectrum antibiotics, along with parenteral nutrition, permanent catheters, chemotherapy and radiotherapy, as well as immunosuppression in patients, is the most important predisposing factors for invasive fungal infections. Fungi are classified according to their morphologies, including yeasts (Cryptococcus spp.), fungi with branched hyphae (Aspergillus spp.), as well as fungi with both morphologies (yeasts and pseudohyphae, as for Candida spp.), which have all been associated with fungal infections in humans.

Fungal biofilms are communities of adherent cells surrounded by an extracellular matrix. These biofilms are commonly found during infection caused by a variety of fungal pathogens. Clinically, biofilm infections can be extremely difficult to eradicate due to their resistance to antifungals and host defenses. Biofilm formation can protect fungal pathogens from many aspects of the innate immune system, including killing by neutrophils and monocytes. Currently, antifungal therapies are scarce and include only four classes of antifungal agents, polyenes, triazoles, echinocandins and flucytosine . The misuse of antifungal agents over the last two decades contributed to antifungal resistance development.Fungal resistance emergence has important clinical implications, as it limits the already small arsenal of antifungal agents, raising the idea of a "post-antifungal" era. Antimicrobial peptides (AMPs) have emerged as new biopharmaceuticals to prevent or treat fungal infections. AMPs are a class of small peptides that widely exist in nature and are an important part of the innate immune system of different organisms. AMPs have a wide range of inhibitory effects against bacteria, fungi, parasites and viruses . Defensins comprise antifungal peptides isolated from various organisms, including plants and mammals . Plant defensins are cationic and have 45-54 amino acids in length. These peptides have typically been isolated from seeds, but can also be found in other plant tissues including leaves, flowers, roots and stems. Most of the plant defensins identified so far have eight cysteine residues that favor structural stability by the formation of four disulfide bonds . In addition, structural studies have shown that plant defensins comprise a triple β-sheet with a parallel helix. Regarding their biological properties, plant defensins have shown activity against bacteria and fungi, both in their planktonic and biofilm modes of growth . Peptides from the cathelicidin family have been isolated from different species of mammals and exhibit broad-spectrum activities against fungi. Cathelicidins are characterized as cationic peptides, consisting of 12-80 amino acids that adopt an α-helix or β-sheet as secondary structures, most of which have 23-37 amino acid residues distributed in amphipathic helices, including LL-37. The activities of LL-37 have been investigated against Candida spp. strains. Human salivary histatins are a group of small histidine-rich proteins constituted from 7 to 38 amino acids first isolated from human parotid saliva. In general, histatins are a multifunctional group of proteins with antimicrobial properties that vary from broad-spectrum to moderate activities. Moreover, histatins have been reported for their effective antifungal activity

ELIGIBILITY:
Inclusion Criteria:

* - Samples obtained from patients with cutaneous fungal infection and systemic fungal infection

Exclusion Criteria:

* Patients diagnosed to be viral or bacterial infections.
* Patients on antibiotic or antifungal treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Samples obtained from patients with cutaneous fungal infection and systemic fungal infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
1.to determine the level at which inhibition of fungi occurs | 6 months
  Determination of defensin ,cathelicidin and histatin is done using broth microdilution method . The procedure involves preparation of twofold dilutions in sterile heart brain broth inside the wells of 96-well microplate.The highest dilution of samples without visible growth after 24 h incubation at 37 °C was considered as minimum inhibitory concentration. . A change in color from blue to pink indicates the growth of bacteria .

SECONDARY OUTCOMES:
measure the percentage of decrease in biofilm formation | 6 month
  The ability of fungal isolates to adhere and to form biofilms in a 96-well plate will be done using the microtiter plate assay.

CONTACTS AND LOCATIONS:
Overall Officials: amal mohamad hosni, lecturer, Study Director — Assiut University; asmaa omar ahmed, assistant professor, Study Chair — Assiut University; mohamad zakaria abd elrahman, professor, Study Chair — Assiut University

REFERENCES:
- [Background] Lionakis MS, Levitz SM. Host Control of Fungal Infections: Lessons from Basic Studies and Human Cohorts. Annu Rev Immunol. 2018 Apr 26;36:157-191. doi: 10.1146/annurev-immunol-042617-053318. Epub 2017 Dec 13. PMID 29237128
- [Background] Chowdhary A, Sharma C, Meis JF. Azole-Resistant Aspergillosis: Epidemiology, Molecular Mechanisms, and Treatment. J Infect Dis. 2017 Aug 15;216(suppl_3):S436-S444. doi: 10.1093/infdis/jix210. PMID 28911045
- [Background] Perlin DS, Rautemaa-Richardson R, Alastruey-Izquierdo A. The global problem of antifungal resistance: prevalence, mechanisms, and management. Lancet Infect Dis. 2017 Dec;17(12):e383-e392. doi: 10.1016/S1473-3099(17)30316-X. Epub 2017 Jul 31. PMID 28774698
- [Background] Huan Y, Kong Q, Mou H, Yi H. Antimicrobial Peptides: Classification, Design, Application and Research Progress in Multiple Fields. Front Microbiol. 2020 Oct 16;11:582779. doi: 10.3389/fmicb.2020.582779. eCollection 2020. PMID 33178164
- [Background] Cools TL, Struyfs C, Drijfhout JW, Kucharikova S, Lobo Romero C, Van Dijck P, Ramada MHS, Bloch C Jr, Cammue BPA, Thevissen K. A Linear 19-Mer Plant Defensin-Derived Peptide Acts Synergistically with Caspofungin against Candida albicans Biofilms. Front Microbiol. 2017 Oct 20;8:2051. doi: 10.3389/fmicb.2017.02051. eCollection 2017. PMID 29104569
- [Background] Oshiro KGN, Rodrigues G, Monges BED, Cardoso MH, Franco OL. Bioactive Peptides Against Fungal Biofilms. Front Microbiol. 2019 Oct 4;10:2169. doi: 10.3389/fmicb.2019.02169. eCollection 2019. PMID 31681179
- [Background] Sathoff AE, Samac DA. Antibacterial Activity of Plant Defensins. Mol Plant Microbe Interact. 2019 May;32(5):507-514. doi: 10.1094/MPMI-08-18-0229-CR. Epub 2019 Mar 29. PMID 30501455
- [Background] Scarsini M, Tomasinsig L, Arzese A, D'Este F, Oro D, Skerlavaj B. Antifungal activity of cathelicidin peptides against planktonic and biofilm cultures of Candida species isolated from vaginal infections. Peptides. 2015 Sep;71:211-21. doi: 10.1016/j.peptides.2015.07.023. Epub 2015 Jul 31. PMID 26238597